CLINICAL TRIAL: NCT06944093
Title: Noninvasive Mechanical Ventilation is Applied to Patients With Hypercapnic Respiratory Failure on the Agitation Scores and Respiratory Parameters
Brief Title: Listen to a Audio Book
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Burak YAVUZ, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/169
Record Dates: First submitted 2025-03-11; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Respiratory Failure With Hypercapnia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Listen to a audio book
  Interventions: Behavioral: audio book
- Control (No Intervention)

INTERVENTIONS:
Behavioral: audio book — Listen to a audio book
  Arms: Experimental

SUMMARY:
This study investigates how listening to audiobooks affects agitation scores and respiratory parameters (like breathing rate, depth, and oxygen saturation) in patients receiving non-invasive mechanical ventilation (NIMV) for hypercapnic respiratory failure in an intensive care unit. Participants will listen to an audiobook of their choice during their 2-hour NIMV treatment. Their agitation levels and respiratory parameters will be measured before, during, and after NIMV application. The goal is to evaluate whether audiobooks can reduce patient agitation and improve respiratory outcomes, offering a low-cost, easy-to-use, and effective approach for better patient care.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 years or older Patients hospitalized in the Chest Diseases Intensive Care Unit Diagnosed with Hypercapnic Respiratory Failure Undergoing Non-invasive Mechanical Ventilation (NIMV) No hearing impairment Conscious and alert patients

Exclusion Criteria:

Patients unwilling to participate or wishing to withdraw from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Agitation Scores | 10 month
Breathing Rate | 10 month
Breathing Depth | 10 month
SpO₂ Levels | 10 month

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk University Faculty of Nursing, Erzurum, Erzurum, Turkey (Türkiye)